CLINICAL TRIAL: NCT00985218
Title: In Vitro Human Embryo Culture System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incept BioSystems, Inc. (Industry)
Responsible Party: Chris Bleck/President and CEO, Incept BioSystems, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBS 001 20080202
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Infertility
Keywords: infertility; embryo development
MeSH Terms: conditions — Infertility | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental arm (Experimental): Embryos cultured in SMART System
  Interventions: Device: SMART System
- Control (Active Comparator): Embryos cultured in microdrops in dishes
  Interventions: Device: Culture dish

INTERVENTIONS:
Device: SMART System — microfluidic embryo culture system
  Other Names: System for Microfluidically-Assisted Reproductive Technology
  Arms: experimental arm
Device: Culture dish — Standard IVF culture dish
  Other Names: dish
  Arms: Control

SUMMARY:
The purpose of this study is to compare the development of human embryos grown in a conventional culture dish to those grown in a new embryo culture device known as the SMART System.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, performance study.

ELIGIBILITY:
Inclusion Criteria - All recruited subjects must meet all of the following inclusion criteria to be enrolled in the study:

1. Female 21 to 35 years of age inclusive
2. First or second IVF cycle
3. Not pregnant
4. No physical abnormalities that would adversely affect oocyte retrieval
5. Male factor is acceptable
6. ICSI is acceptable
7. 10 zygotes or more

Exclusion Criteria- Potential subjects are excluded from the study if any of the following conditions exist:

1. The sperm were retrieved using TESE or MESA
2. The embryos were created with either donor oocytes or donor sperm.
3. Medical condition precluding a safe pregnancy
4. Medical condition disqualifying the subject from safely participating in the study in the judgment of the investigator

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
rate of development of human embryos | Day 3 (t=72 hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Pool, Ph.D., HCLD, Principal Investigator — Fertility Center of San Antonio; Joseph Conaghan, Ph.D., HCLD, Principal Investigator — Pacific Fertility Center; Rodney Wade, BSA, MS, ELD, Principal Investigator — Southeastern Fertility Center; Kelvin L Fry, B. SC., Principal Investigator — Florida Fertility Institute
Locations (4):
- United States (4):
  - Pacific Fertility Center, San Francisco, California
  - Florida Fertility Institute, Clearwater, Florida
  - Southeastern Fertility Center, Mt. Pleasant, South Carolina
  - Fertility Center of San Antonio, San Antonio, Texas